CLINICAL TRIAL: NCT05693415
Title: Primary Osteoarthritis Lumbar Spine Presenting as Chronic Low Back Pain or Sciatica or Both (Prolapsed Lumbar Disc Syndrome): Establishing Its Cause, Pathogenesis and Treatment.
Brief Title: Primary Osteoarthritis Lumbar Spine: Establishing Its Cause, Pathogenesis and Treatment.
Status: Completed | Type: Observational
Sponsor: Knee Pain Clinic (Other)
Responsible Party: Principal Investigator, DR R C Agrawal, Principal Investigator, Knee Pain Clinic
Other Study IDs: 1002
Record Dates: First submitted 2022-10-26; First posted 2023-01-23 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Lumbar Osteoarthritis
Keywords: Osteoarthritis; Lumbar Spine; Intervertebral Joint; Capsule Contracture; Discectomy; Ideopathic
MeSH Terms: conditions — Osteoarthritis, Spine; Osteoarthritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control Group: No treatment
- Trial Group: Non drug and none surgical treatment of contracted Lumber Spine
  Other Names:
  Contracture Correction Therapy

SUMMARY:
The study was about a root cause of Primary Osteoarthritis Lumbar Spine producing disabilities in sitting, climbing and walking etc. In advance stage the person is bereft of his/her personal physical activities. The prevalent treatment is temporary and dis-satisfactory. A new treatment was designed and a trial was conducted on 154 patients (100 in the trial group, 50 in the control group) for a duration of six months.

DETAILED DESCRIPTION:
The study was focused on establishing the cause, pathogenesis and treatment of painful Lumbar Spine disease (Primary Osteoarthritis Lumbar Spine = OA Lumbar Spine) at present the exact cause and treatment are not known. It was aimed to find out to latter through a hypothesis by designing a treatment and testing it with a clinical trial.

This established that the deficient full extension of the spinal joints (intervertebral joints between the adjacent vertebrae from T12 to S1) producing contracture in their capsules in front, was the cause and the correction (Contracture Correction Therapy = CCT) was the cure of the disease. The correction was carried out by intermittent and sustained extension of the lumbar spin through three designed body postures.

ELIGIBILITY:
Inclusion Criteria:

* Age =>30 and <=90 years
* Back/leg pain or both combined, which appears without any apparent cause, exacerbated by exertion and subsides by rest.
* Presence of limited morning stiffness
* No history of infection, inflammation or trauma to rule out secondary OA
* Disability in sitting, climbing stairs or walking

Exclusion Criteria:

* Neckache
* Frozen shoulder
* Central obesity
* Acute Lumbago
* X-ray spine with no OA signs

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Group includes people across locations in and Gwalior city. Trial was based on "Pragmatic Cluster Randomized Controlled Trial", also known as Cluster Randomized Trial (CRT) or Group Randomized Trial. In this variety pre-existing groups, called clusters, of individuals are randomly allocated to treatment arms. The subjects, who consulted me, were of two types. The type I wanted to avoid surgery, had tried other nonsurgical options and did not want those anymore. These patients were included in trial group and took my designed treatment (Contracture Correction Therapy = CCT). The other type of patients who did not consent for the new treatment were included in the control group.
Sampling Method: Non-Probability Sample
Enrollment: 154 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-10-15 (Actual)

PRIMARY OUTCOMES:
The Western Ontario and McMaster Universities Arthritis Index (WOMAC) | Change from baseline The Western Ontario and McMaster Universities Arthritis Index Osteoarthritis score at 6, 12, 24 weeks
  It is a self-administered questionnaire consisting of 24 items divided into 3 subscales

SECONDARY OUTCOMES:
Oswestry Disability Index | Change from baseline Oswestry Disability Index score at 6, 12, 24 weeks
  Patient-completed questionnaire which gives a subjective percentage score of level of function (disability) in activities of daily living in those rehabilitating from low back pain.
EuroQol Visual Analogue Scale score | Change from baseline EuroQol Visual Analogue Scale score at 6, 12, 24 weeks
  The EQ-VAS is a vertical visual analogue scale that takes values between 100 (best imaginable health) and 0 (worst imaginable health), on which patients provide a global assessment of their health.

CONTACTS AND LOCATIONS:
Overall Officials: R C Agrawal, MS Surgery, Principal Investigator — Knee Pain Clinic
Locations (6):
- India (6):
  - Arogya Sadan Nursing Home, Bhind, Madhya Pradesh
  - Sai Baba Dharmarth Chikitsalaya, Gwalior, Madhya Pradesh
  - Knee Pain Clinic, Gwalior, Madhya Pradesh
  - Lok Hitkari Trust Health Camp, Gwalior, Madhya Pradesh
  - Parashar Poly Clinic, Gwalior, Madhya Pradesh
  - Dr. Shukla Surgery Center, Morena, Madhya Pradesh

IPD SHARING:
Plan to Share IPD: No